CLINICAL TRIAL: NCT00480324
Title: Efficacy, Safety, Reactogenicity and Immunogenicity Study of the Lyophilised Formulation of Rotarix Vaccine in Healthy Japanese Infants
Brief Title: Efficacy, Safety, Reactogenicity & Immunogenicity of the Rotarix Vaccine in Japanese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 107625; 2015-001543-36 (EudraCT Number)
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rotarix Group (Experimental): Subjects received 2 oral doses of Rotarix according to a 0, 1 month schedule.
  Interventions: Biological: Rotarix
- Placebo Group (Placebo Comparator): Subjects received 2 oral doses of placebo according to a 0, 1 month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix — Two-dose oral vaccination.
  Arms: Rotarix Group
Biological: Placebo — Two-dose oral administration.
  Arms: Placebo Group

SUMMARY:
This study is undertaken to provide the regulatory authorities in Japan with immunogenicity, efficacy, safety and reactogenicity data of GSK Biologicals' Human Rotavirus [HRV] vaccine, given as a 2-dose primary vaccination, in healthy Japanese infants aged approximately 2 months at the time of the first dose and previously uninfected with HRV. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Combined diphtheria and tetanus toxoids and acellular pertussis (DTPa) and Hepatitis B (HBV) vaccines are allowed to be co-administered along with Rotarix vaccine/Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infant between, and including, 6 and 14 weeks (42-104 days) of age at the time of the first vaccination.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Born between a gestation period of 36 and 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the HRV vaccine within 30 days preceding the first dose of HRV vaccine, or planned use during the study period.
* History of use of experimental rotavirus vaccine.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for intussusception.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition determined by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Previous confirmed occurrence of RV GE.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* A family history of congenital or hereditary immunodeficiency.
* Acute disease at the time of enrolment.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 765 (Actual)
Dates: Start 2007-06-19 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Japan (13):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=272

REFERENCES:
- [Background] Kawamura N, Tokoeda Y, Oshima M, Okahata H, Tsutsumi H, Van Doorn LJ, Muto H, Smolenov I, Suryakiran PV, Han HH. Efficacy, safety and immunogenicity of RIX4414 in Japanese infants during the first two years of life. Vaccine. 2011 Aug 26;29(37):6335-41. doi: 10.1016/j.vaccine.2011.05.017. Epub 2011 Jun 2. PMID 21640780
- [Background] Kawamura N et al. Efficacy of Human Rotavirus (G1P[8] strain) Vaccine (HRV) RIX4414 in Japanese Infants during the Two-year Efficacy Follow-up Period. Abstract presented at the 114th Annual Meeting of Japan Pediatric Society (JPS). Tokyo, Japan, 12-14 August 2011.
- [Background] Kawamura N et al. Efficacy of human rotavirus vaccine RIX4414 in Japanese infants from 2 weeks post dose 2 up to data lock point. Abstract presented at the 28th meeting of European Society for Paediatric Infectious Diseases (ESPID). Nice, France, 4-8 May 2010.
- [Background] Buyse H, Vinals C, Karkada N, Han HH. The human rotavirus vaccine Rotarix in infants: an integrated analysis of safety and reactogenicity. Hum Vaccin Immunother. 2014;10(1):19-24. doi: 10.4161/hv.26476. Epub 2013 Oct 8. PMID 24047799
- [Derived] Bergman H, Henschke N, Hungerford D, Pitan F, Ndwandwe D, Cunliffe N, Soares-Weiser K. Vaccines for preventing rotavirus diarrhoea: vaccines in use. Cochrane Database Syst Rev. 2021 Nov 17;11(11):CD008521. doi: 10.1002/14651858.CD008521.pub6. PMID 34788488
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 508 | 257
Completed | 476 | 241
Not Completed | 32 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 14 | 5
Not completed — Lost to Follow-up | 17 | 8
Not completed — Subject's mother pregnant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 508 | 257 | 765
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 7.7 (1.99) | 7.7 (2.05) | 7.7 (2.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 134 | 363
  Male | 279 | 123 | 402

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Rotavirus (RV) Gastroenteritis (GE) Leading to Medical Intervention and Caused by the Circulating Wild-type RV Strains
Description: Rotavirus (RV) gastroenteritis (GE) was defined as an episode of any severity GE leading to a medical intervention occurring at least two weeks after dose 2 in which rotavirus other than vaccine strain is identified in a stool sample collected as soon as possible but preferably not later than 7 days after the start of the episode.
Time Frame: From 2 weeks after Dose 2 up to 2 years of age
Population: The analysis was performed on the according-to-protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 498 | 250
subjects | 14 | 34

2. Secondary Outcome: Number of Subjects Reporting Severe Rotavirus (RV) Gastroenteritis (GE) Leading to Medical Intervention and Caused by the Circulating Wild-type RV Strains
Description: A subject was considered as reporting severe rotavirus gastroenteritis when the subject scored 11 or more on a 20-point scoring system (Vesikari scoring system).
Time Frame: From 2 weeks after Dose 2 up to 2 years of age
Population: The analysis was performed on the according-to-protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 498 | 250
subjects | 2 | 12

3. Secondary Outcome: Number of Subjects Reporting Any Rotavirus (RV) Gastroenteritis (GE) and Severe RV GE Leading to Medical Intervention and Caused by the Circulating Wild-type RV Strains of G1 Type
Description: Rotavirus (RV) gastroenteritis (GE) was defined as an episode of any severity GE leading to a medical intervention occurring at least two weeks after dose 2 in which rotavirus other than vaccine strain is identified in a stool sample collected as soon as possible but preferably not later than 7 days after the start of the episode.
  Severe RV GE was defined as an episode of rotavirus gastroenteritis with score ≥ 11 on a 20-point scoring system (Vesikari scoring system).
Time Frame: From 2 weeks after Dose 2 up to 2 years of age
Population: The analysis was performed on the according-to-protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 498 | 250
subjects
  Any RV GE | 4 | 13
  Severe RV GE | 1 | 6

4. Secondary Outcome: Number of Subjects Reporting Any Rotavirus (RV) Gastroenteritis (GE) and Severe RV GE Leading to Medical Intervention and Caused by the Circulating Wild-type RV Strains of Non-G1 Types
Description: Rotavirus (RV) gastroenteritis (GE) was defined as an episode of any severity GE leading to a medical intervention occurring at least two weeks after dose 2 in which rotavirus other than vaccine strain is identified in a stool sample collected as soon as possible but preferably not later than 7 days after the start of the episode.
  Severe rotavirus gastroenteritis was defined as an episode of rotavirus gastroenteritis with score ≥ 11 on a 20-point scoring system (Vesikari scoring system).
Time Frame: From 2 weeks after Dose 2 up to 2 years of age
Population: The analysis was performed on the according-to-protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 498 | 250
subjects
  Any RV GE | 10 | 21
  Severe RV GE | 1 | 6

5. Secondary Outcome: Number of Subjects Hospitalized Due to Rotavirus (RV) Gastroenteritis (GE) Caused by the Circulating Wild-type RV Strains
Description: as for outcome 1
Time Frame: From 2 weeks after Dose 2 up to 2 years of age
Population: The analysis was performed on the according-to-protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 498 | 250
subjects | 1 | 2

6. Secondary Outcome: Number of Subjects Reporting Any Rotavirus (RV) Gatroenteritis (GE) and Severe RV GE Leading to Medical Intervention and Caused by the Circulating Wild-type RV Strains
Description: as for outcome 4
Time Frame: From Dose 1 up to 2 years of age
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 257
subjects
  Any RV GE | 14 | 36
  Severe RV GE | 2 | 13

7. Secondary Outcome: Serum Anti-rotavirus Immunoglobulin A (IgA) Antibody Concentration
Description: Anti-rotavirus immunoglobulin A antibody concentrations are given as geometric mean concentrations (GMCs). Arbitrary 'zero' values were set in the Placebo Group since the GMC was below the assay cut-off value (20 U/mL).
Time Frame: 2 months after Dose 2
Population: The analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 34 | 20
Units per milliliter (U/mL) | 217.0 [109.9 to 428.6] | 0 [0 to 0]

8. Secondary Outcome: Number of Subjects Seroconverted for Anti-rotavirus Immunoglobulin A (IgA) Antibodies
Description: Seroconversion was defined as the appearance of anti-rotavirus immunoglobulin A antibody concentration ≥ 20 units (U)/milliliter (mL) in subjects initially (i.e. prior to the first dose of rotarix) seronegative.
Time Frame: 2 months after Dose 2
Population: The analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 34 | 20
subjects | 29 | 1

9. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited symptoms assessed include cough, diarrhoea, fever, irritability, loss of appetite and vomiting.
Time Frame: During the 8-day follow-up period after each dose
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 257
subjects
  Cough | 184 | 92
  Diarrhoea | 43 | 14
  Fever | 62 | 22
  Irritability | 261 | 125
  Loss of appetite | 81 | 33
  Vomiting | 74 | 36

10. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day follow-up period after each dose
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 257
subjects | 279 | 144

11. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to 2 years of age
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 257
subjects | 72 | 44

ADVERSE EVENTS:
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 72/508 | 44/257
Other Adverse Events (participants affected / at risk) | 411/508 | 204/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=508) | Placebo Group (N=257)
Pneumonia (Infections and infestations) | 12 | 4
Bronchitis (Infections and infestations) | 14 | 0
Gastroenteritis (Infections and infestations) | 11 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pharyngitis (Infections and infestations) | 5 | 3
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 6 | 2
Respiratory syncytial virus infection (Infections and infestations) | 5 | 3
Exanthema subitum (Infections and infestations) | 3 | 2
Febrile convulsion (Nervous system disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Bronchopneumonia (Infections and infestations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Otitis media acute (Infections and infestations) | 1 | 3
Pyrexia (General disorders) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Convulsion (Nervous system disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 2
Influenza (Infections and infestations) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Acute tonsilitis (Infections and infestations) | 1 | 1
Adenovirus infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 2
Enterocolitis viral (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Kawasaki's disease (Vascular disorders) | 1 | 1
Laryngitis (Infections and infestations) | 2 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=508) | Placebo Group (N=257)
Eczema (Skin and subcutaneous tissue disorders) | 72 | 29
Upper respiratory tract infection (Infections and infestations) | 50 | 25
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 33 | 16
Nasopharyngitis (Infections and infestations) | 31 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 21
Cough (General disorders) | 184 | 92
Diarrhoea (General disorders) | 43 | 14
Fever (General disorders) | 62 | 22
Irritability (General disorders) | 261 | 125
Loss of appetite (General disorders) | 81 | 33
Vomiting (General disorders) | 74 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.